CLINICAL TRIAL: NCT07108127
Title: Phase II Clinical Study on the Efficacy and Safety of Trastuzumab Biosimilars and Pertuzumab Biosimilars Combined With Chemotherapy for Neoadjuvant Treatment of Patients With Locally Advanced HER2-positive Rectal Cancer
Brief Title: Efficacy and Safety of Trastuzumab Biosimilars and Pertuzumab Biosimilars Combined With Chemotherapy for Neoadjuvant Treatment of Patients With Locally Advanced HER2-positive Rectal Cancer
Acronym: NePHera
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K7720; 2024-PUMCH-E-013 (Other: Peking Union Medical College Hospital)
Record Dates: First submitted 2025-03-25; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer; HER2-positive
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX

STUDY DESIGN:
Intervention Model Description: Trastuzumab biosimilars and pertuzumab biosimilars in combination with oxaliplatin and capecitabine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Trastuzumab biosimilars and pertuzumab biosimilars in combination with oxaliplatin and capecitabine
  Interventions: Drug: Trastuzumab biosimilars and pertuzumab biosimilars plus XELOX

INTERVENTIONS:
Drug: Trastuzumab biosimilars and pertuzumab biosimilars plus XELOX — Trastuzumab biosimilars and pertuzumab biosimilars combined with oxaliplatin and capecitabine

SUMMARY:
The purpose of this study was to evaluate the complete response rate (CR) of trastuzumab biosimilars and pertuzumab biosimilars combined with oxaliplatin and capecitabine in neoadjuvant treatment of patients with locally advanced (cT3/T4, N+, distance from the lower edge of the tumor to the anal verge ≤12 cm) HER2-positive rectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Patients with rectal cancer confirmed by histology or cytology; locally advanced (cT3/T4, N+, distance from the lower edge of the tumor to the anal verge ≤ 12 cm) rectal adenocarcinoma (using the 8th edition of the AJCC TNM staging);
3. HER2 positive after detection: HER2 positive is defined as IHC test result 3+, or IHC test result 2+ and FISH method confirms positive HER2 gene amplification;
4. Tumor tissue gene test RAS/BRAF is wild type (previous test results are acceptable);
5. Previous treatment meets the following requirements: no previous anti-tumor treatment;
6. ECOG PS score 0-1;
7. Expected survival period of at least 3 months;
8. Adequate organ function, laboratory tests meet the following criteria (no blood transfusion or hematopoietic stimulating factor treatment within 14 days):

   1. Absolute neutrophil count (ANC) ≥ 1.5×109/L
   2. Hemoglobin (Hb) ≥ 90g/L
   3. Platelets ≥ 100×109/L
   4. Albumin ≥ 30g/L
   5. Serum creatinine ≤ 1.5×ULN and creatinine clearance > 50 mL/min (calculated according to Cockcroft-Gault formula)
   6. Total bilirubin ≤ 1.5×ULN;
   7. Alanine aminotransferase, aspartate aminotransferase ≤ 2.5×ULN, alanine aminotransferase, aspartate aminotransferase ≤ 5×ULN for patients with liver metastasis;
   8. Activated partial thromboplastin time ≤ 1.5×ULN; international normalized ratio ≤ 1.5×ULN.
9. Eligible individuals (male and female) of childbearing potential must agree to use reliable contraceptive methods (hormonal contraceptives, barrier methods or abstinence) with their partners during the trial and for at least 6 months after the last dose. Female individuals of childbearing age must have a negative blood pregnancy test within 7 days before enrollment;
10. Fully understand this clinical trial and voluntarily sign a written informed consent.

Exclusion Criteria:

1. Patients who have received anti-HER2 drug treatment in the past;
2. Patients with known clinical symptoms of central nervous system metastasis or meningeal metastasis, or other evidence that individual central nervous system metastasis or meningeal metastasis has not been controlled, and are judged by the investigator to be unsuitable for inclusion;
3. Patients who are receiving long-term immunosuppressive therapy (such as cyclosporine) or require daily systemic steroid therapy (such as >20 mg prednisone or equivalent drugs), except those who use local glucocorticoids by nasal spray, inhalation or other routes;
4. The adverse reactions of previous anti-tumor treatment have not recovered to CTCAE 5.0 grade evaluation ≤1 (except for toxicities such as alopecia that the investigator judges to have no safety risks);
5. Clinically significant gastrointestinal diseases, including but not limited to severe liver disease, malabsorption syndrome, ulcerative colitis, inflammatory bowel disease;
6. Peripheral neuropathy of grade 3 or above;
7. Known low level or deficiency of dihydropyrimidine dehydrogenase (DPD);
8. Individuals who have undergone major surgery or invasive intervention within 28 days before the first dose (excluding puncture biopsy, central venous catheter chemotherapy, infusion port, stent implantation and bile duct drainage for relieving biliary obstruction, and cholecystostomy surgery);
9. Participating in another clinical trial at the same time;
10. Using any Chinese herbal medicine or Chinese patent medicine with anti-cancer activity approved by the State Food and Drug Administration within 14 days before the first dose (regardless of the type of cancer);
11. Known to have severe allergic reactions to the study drug or other ingredients or excipients in the preparation;
12. Active bacterial, fungal or viral infection within 14 days before the first dose (defined as requiring intravenous antibacterial, antifungal or antiviral drug treatment). Individuals who have no clinical manifestations of active infection before the first dose and are given preventive treatment for infection may be considered for inclusion in the group;
13. Within 7 days before the first dose, there is uncontrolled serous effusion that requires frequent drainage or medical intervention (such as pleural effusion, peritoneal effusion, pericardial effusion, etc., which requires additional intervention within 2 weeks after intervention, excluding exfoliative cytology testing of exudate);
14. Suffering from autoimmune diseases, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis), autoimmune hepatitis, systemic sclerosis (scleroderma, etc.), Hashimoto's thyroiditis (exceptions are shown below), autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome), etc. The following conditions are excluded: type 1 diabetes, hypothyroidism that is stable with hormone replacement therapy (including hypothyroidism caused by autoimmune thyroid disease), psoriasis or vitiligo that does not require systemic treatment;
15. HBsAg positive and HBV-DNA higher than the measurable lower limit or 1000 copies/mL (500 IU/mL) (whichever is lower), HCV antibody positive and HCV-RNA higher than the measurable lower limit or 1000 copies/mL (whichever is lower); HIV antibody test positive;
16. History of non-infectious interstitial lung disease, or interstitial pneumonia requiring hormone treatment;
17. History of severe cardiovascular disease, including but not limited to:

    1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block, etc.;
    2. QTcF > 450 milliseconds at rest (if the first 12-lead electrocardiogram QTcF > 450 milliseconds, can be repeated twice, take the average of 3 times);
    3. Acute coronary syndrome, congestive heart failure, heart or other vascular stent implantation, angioplasty or cardiac surgery, stroke or other cardiovascular events of grade 3 or above within 6 months before the first administration;
    4. New York Heart Association heart function grade ≥ II or left ventricular ejection fraction <50%;
    5. Any factors that increase the risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death of first-degree relatives under 40 years old, use of any concomitant drugs known to prolong the QT interval;
    6. Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg during the screening period). 18) History of other malignant tumors within 5 years or other active malignant tumors at the same time (cured localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc. can be included);

19) Vaccinated with live vaccine within 28 days before randomization. Note: Seasonal influenza vaccine is an inactivated vaccine in a broad sense and is allowed to be used; intranasal influenza vaccine is a live vaccine and is not allowed to be used (applicable to immunotherapy); 20) Known mismatch repair protein deficiency (dMMR) or microsatellite high instability (MSI-H) 21) Current psychiatric disorders that affect compliance; 22) Pregnant or lactating women; 23) Patients who have used strong CYP3A4 inhibitors or strong inducers, or strong UGT1A1 inhibitors within 2 weeks before the first dose (applicable to FOLFIRI regimen treatment); 24) The investigator believes that the patient is not suitable for participating in this clinical trial for other reasons, including but not limited to: patients with concurrent serious or uncontrollable medical conditions, safety risks, interference with the interpretation of research results, and impact on trial compliance, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CR | through study completion, an average of 1 year
  Complete remission (CR) including pCR and cCR

SECONDARY OUTCOMES:
ORR | through study completion, an average of 1 year
  overall response rate
DFS | through study completion, an average of 1 year
  disease free survival
R0 resection rate | through study completion, an average of 1 year
  R0 resection rate
TRG | through study completion, an average of 1 year
  tumor regression grade

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China